CLINICAL TRIAL: NCT03795519
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Olinciguat ([14C]-IW-1701) Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Trial to Study the Absorption, Metabolism, and Excretion of [14C]-Olinciguat in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OLI-103
Record Dates: First submitted 2018-12-14; First posted 2019-01-07 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Male Volunteers (Experimental): Single oral dose of [14C]-olinciguat
  Interventions: Drug: [14C]-olinciguat

INTERVENTIONS:
Drug: [14C]-olinciguat — oral capsule
  Other Names: 14C-IW-1701

SUMMARY:
The primary objective is to characterize the pharmacokinetics (PK) of olinciguat and total radioactivity and to assess the elimination of total radioactivity from a single oral dose of [14C]-olinciguat.

DETAILED DESCRIPTION:
OLI-103 is a Phase 1 open-label, nonrandomized, single-dose study in up to 8 subjects that will be conducted at a single center in the US. Safety assessments will be performed throughout the clinic period and multiple PK samples will be collected. Subjects will be confined to the clinical research center for at least 8 days.

The purpose of the study is to determine the absorption, metabolism, and excretion of [14C]-olinciguat and to characterize and determine, where possible, the metabolites present in plasma, urine, and feces after a single oral dose. The study will help identify and characterize olinciguat metabolites, evaluate the likelihood of effects of liver or kidney impairment on the disposition of olinciguat, and assess the likelihood of drug-drug interactions with olinciguat.

ELIGIBILITY:
Inclusion Criteria:

* Males of any race, between 18 and 55 years of age, inclusive
* Body mass index between 18 and 32 kg/m2, inclusive
* Subject is in good health and has no clinically significant findings on physical examination
* Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and for at least 90 days after the final dose of study drug

Exclusion Criteria:

* Any active or unstable clinically significant medical condition
* Use of any prescribed or non-prescribed medication

Additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Amount of total radioactivity excreted in urine (Aeu) and feces (Aef) | up to Day 15
Cumulative Aeu and cumulative Aef | up to Day 15
Percentage of total radioactivity excreted in urine (feu) and feces (fef) | up to Day 15
Cumulative feu and cumulative fef | up to Day 15
Percentage of total radioactivity in total excreta (feces + urine) | up to Day 15
Area under the concentration-time curve (AUC) from time zero to infinity (AUC0-inf) of olinciguat in plasma | up to Day 15
AUC0-inf of total radioactivity in plasma and whole blood | up to Day 15
AUC from time zero to the last quantifiable concentration (AUC0-last) of olinciguat in plasma | up to Day 15
AUC0-last of total radioactivity in plasma and whole blood | up to Day 15
Maximum observed concentration (Cmax) of olinciguat in plasma | up to Day 15
Cmax of total radioactivity in plasma and whole blood | up to Day 15
Time of Cmax (Tmax) of olinciguat in plasma | up to Day 15
Tmax of total radioactivity in plasma and whole blood | up to Day 15
Apparent terminal elimination half-life (t1/2) of olinciguat in plasma | up to Day 15
t1/2 total radioactivity in plasma and whole blood | up to Day 15
Apparent total clearance of olinciguat (CL/F) | up to Day 15
Apparent volume of distribution of olinciguat (Vz/F) | up to Day 15
AUC0-inf of plasma olinciguat concentration relative to AUC0-inf of plasma total radioactivity (AUC0-inf Ratio of Plasma Olinciguat/Plasma Total Radioactivity) | up to Day 15
AUC0-inf of whole blood total radioactivity to AUC0-inf of plasma total radioactivity (AUC0-inf Ratio of Blood Total Radioactivity/Plasma Total Radioactivity) | up to Day 15

SECONDARY OUTCOMES:
Levels of metabolite radioactivity excreted in urine and feces | up to Day 15
AUC0-inf of metabolite radioactivity levels in plasma | up to Day 15
AUC0-inf of plasma metabolite radioactivity levels relative to AUC0-inf of plasma total radioactivity (Plasma AUC0-inf Ratio of Metabolite Radioactivity/Total Radioactivity) | up to Day 15
Chromatographic retention time of metabolites | up to Day 15
Molecular ion mass of metabolites | up to Day 15
Characteristic mass spectrometry fragmentation ions of metabolites | up to Day 15
Chemical structures (graphical representations showing atom connectivity) proposed for plasma, urine, and feces metabolites | up to Day 15
Number(s) of participants with ≥1 treatment-emergent serious adverse event (SAE) | up to Day 15
Number(s) of participants with ≥1 adverse event (AE) leading to study drug discontinuation | up to Day 15
Number(s) of participants with ≥1 Grade ≥3 AE (per CTCAE v. 5.0) | up to Day 15
Number(s) of participants with ≥1 clinically significant abnormal physical examination finding | up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Bina Tejura, MD, Study Director — Ironwood Pharmaceuticals, Inc.
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No